CLINICAL TRIAL: NCT05972382
Title: Investigating Associations Between Neck Flexor Muscle Fatigue, Cervical Joint Position Sense Errors, and Headache Pain and Disability in Individuals With Chronic Cervicogenic Headache
Brief Title: Associations Between Neck Muscle Fatigue, Joint Position Sense, and Headache in Cervicogenic Headache
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: CGH01
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervicogenic Headache: Individuals with chronic cervicogenic headache (>3 months duration)
  Interventions: Diagnostic Test: Quantitative Sensory and Neurophysiological Testing

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory and Neurophysiological Testing — Participants will undergo the following quantitative sensory and neurophysiological diagnostic tests:
  Surface electromyography (EMG) of the neck flexor muscles during the craniocervical flexion test to assess neck flexor muscle fatigue. EMG sensors will be placed over the sternocleidomastoid and longus colli muscles. Cervical joint position error testing to evaluate proprioceptive awareness and cervicocephalic kinesthetic sensibility. Participants will be seated upright and blindfolded.

SUMMARY:
This research study aims to better understand the relationships between neck muscle function, neck joint position sense, and headache pain and disability in people with chronic cervicogenic headache. Cervicogenic headache is headache originating from the neck area.

Participants will fill out questionnaires about their headache pain and ability to do daily activities. They will also do tests to measure neck muscle fatigue and neck joint position sense. Researchers will analyze if those with more neck muscle fatigue and poorer joint position sense have worse headache pain and disability.

The results may improve understanding of cervical spine factors related to cervicogenic headache. This could help guide more targeted treatment approaches.

DETAILED DESCRIPTION:
Chronic cervicogenic headache (CGH) is characterized by chronic headache originating from the upper cervical spine and occipital region. CGH is associated with impairments in cervical muscular control and proprioception or joint position sense. However, relationships between these cervical impairments and headache symptoms are not fully elucidated.

This cross-sectional quantitative study aims to investigate associations between neck flexor muscle fatigue, cervical joint position sense, and clinical headache parameters like pain and disability in individuals with CGH.

A sample of 30 adults ages 18-65 years old with CGH longer than 3 months duration and more than 15 headache days per month will be recruited from neurology clinics. Participants will attend a single 2 hour study visit.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 years
* Chronic CGH (>3 months duration)
* Headache frequency ≥15 days/month

Exclusion Criteria:

* Cervical nerve root compression or other specific pathologies explaining headache
* History of cervical spine surgery
* Botulinum toxin injections in cervical musculature in past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with chronic cervicogenic headache recruited from neurology clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Headache Pain Intensity | Baseline
  Average headache pain over the past week rated on a 0-10 Numerical Rating Scale (NRS). Participants asked to rate their average pain level over the past week on a 0 to 10 scale, where 0 is no pain and 10 is the worst possible pain.

SECONDARY OUTCOMES:
Headache Disability | Baseline
  Total score on the 25-item Headache Disability Inventory (HDI) questionnaire, assessing headache-related disability over the past month. Each item scored as yes (4 points), sometimes (2 points), or no (0 points). Total score ranges from 0 to 100, with higher scores indicating greater disability.
Neck Flexor Fatigue | baseline
  Change in mean surface electromyography (EMG) amplitude (measured in microvolts) of the sternocleidomastoid and longus colli muscles from start to end of a 30-second craniocervical flexion contraction at 50% maximum voluntary contraction (MVC).
Cervical Joint Position Sense | Baseline
  Absolute error in degrees between perceived and actual head repositioning after returning from 20 degrees of active right cervical rotation. Average error over 3 trials used.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No